CLINICAL TRIAL: NCT05083390
Title: Double-blind, Randomised, Placebo-controlled, Phase IIb Trial on the Efficacy and Safety of Norursodeoxycholic Acid Tablets in Patients With Non-alcoholic Steatohepatitis (NASH)
Brief Title: Norursodeoxycholic Acid vs. Placebo in NASH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dr. Falk Pharma GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NUT-3/NAS
Record Dates: First submitted 2021-10-06; First posted 2021-10-19 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Nonalcoholic Steatohepatitis
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — 24-norursodeoxycholic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- norUrsodeoxycholic acid 1500 mg/day (Experimental): 3 film-coated tablets once daily for 72 weeks containing in total norUrsodeoxycholic acid 1500 mg
  Interventions: Drug: norUrsodeoxycholic acid
- norUrsodeoxycholic acid 1000 mg/day (Experimental): 3 film-coated tablets once daily for 72 weeks containing in total norUrsodeoxycholic acid 1000 mg
  Interventions: Drug: norUrsodeoxycholic acid
- Placebo to norUrsodeoxycholic acid (Placebo Comparator): 3 film-coated tablets once daily for 72 weeks containing placebo to norUrsodeoxycholic acid
  Interventions: Drug: norUrsodeoxycholic acid

INTERVENTIONS:
Drug: norUrsodeoxycholic acid — 500 mg norUrsodeoxycholic acid or placebo film-coated tablets; 3 tablets/day
  Other Names: norucholic acid; norUDCA; NCA

SUMMARY:
This is a double-blind, randomised, multi-centre, placebo-controlled, comparative, phase IIb trial. The trial will be conducted with three treatment groups in the form of a parallel group comparison and will serve to compare oral treatment with either 1500 mg/d or 1000 mg/d norUDCA tablets vs. placebo tablets for the treatment of NASH.

ELIGIBILITY:
Inclusion Criteria:

* Must be willing to participate in the study and provide written informed consent
* Male or female patients ≥ 18 and < 75 years
* Centrally assessed histological evidence of NASH and liver fibrosis
* Women of childbearing potential agree to use a highly effective method of birth control during the entire duration of the trial and for 4 weeks following the last dose of trial treatment

Exclusion Criteria:

* Patients taking prohibited medications
* Presence of liver cirrhosis
* Type 1 diabetes or uncontrolled Type 2 diabetes
* History or presence of any other significant concomitant liver diseases
* History of liver transplantation
* BMI >45 kg/m^2
* Any known relevant infectious disease (e.g., active tuberculosis, acquired immunodeficiency syndrome [AIDS]-defining diseases)
* Abnormal renal function (glomerular filtration rate estimated from cystatin C < 30 ml/min) at screening visit
* Any active malignant disease (except for basal cell carcinoma)
* Existing or intended pregnancy or breast-feeding

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Number of participants with resolution of NASH, assessed by centrally scored liver histology, and no worsening of fibrosis AND/OR improvement of fibrosis, and no worsening of NAS | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Trauner, MD, Principal Investigator — Medical University of Vienna, Department of Internal Medicine III
Locations (1):
- Medical University of Vienna, Department of Internal Medicine III, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
It is not yet decided which data will be made available. Neither a time frame can be indicated yet.